CLINICAL TRIAL: NCT07280728
Title: Effectiveness of a Nurse-Led Face-to-Face Educational Intervention on Clinical Stability, Compliance, and Self-Care in Patients With Heart Failure Three Months After Hospital Discharge: An Open-Label Randomized Controlled Trial (EDUCATE Study)
Brief Title: Nurse-Led Education for Heart Failure Self-Care and Stability
Acronym: EDUCATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale di Lodi (Other)
Responsible Party: Principal Investigator, Greta Ghizzardi, Nurse Researcher, Azienda Socio Sanitaria Territoriale di Lodi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDUCATE Study; CET 195-2025 (Registry Identifier: registro dei pareri del CET Lombardia 1)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Heart Failure
Keywords: Heart Failure; Self-Care; Patient Education; Nurse-Led Intervention; Teach-Back; Clinical Stability; Medication Adherence; Randomized Controlled Trial; Post-Discharge Care
MeSH Terms: conditions — Heart Failure; Medication Adherence

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, randomized controlled trial with a 1:1 allocation ratio. Participants will be assigned to either the intervention group, receiving a structured nurse-led educational session using the teach-back method, or the control group, receiving standard follow-up care. Outcomes will be assessed at 3, 6, 9, and 12 months after enrollment.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-Led Face-to-Face Educational Intervention (Experimental): Participants in this arm will receive a structured 30-minute educational session conducted by trained nurses during the first outpatient cardiology visit, approximately 30 days after hospital discharge. The session includes symptom assessment, individualized education using the teach-back method, and delivery of educational materials developed by Penn Nursing Science. A reinforcement phone call will be made one month later, and the educational session will be repeated at six months.
  Interventions: Behavioral: Nurse-Led Face-to-Face Educational Intervention (Teach-Back Method)
- Standard Follow-Up Care (No Intervention): Participants in this arm will receive standard follow-up care, consisting of a 15-minute telephone contact one week after the first outpatient cardiology visit and monthly phone calls thereafter until 12 months post-discharge. During each call, nurses will reinforce medication adherence and collect basic clinical parameters such as blood pressure, heart rate, and weight.

INTERVENTIONS:
Behavioral: Nurse-Led Face-to-Face Educational Intervention (Teach-Back Method) — A 30-minute structured educational session delivered by trained nurses during the first outpatient cardiology visit (about 30 days after discharge). The intervention includes symptom assessment, individualized education using the teach-back method, and delivery of educational materials from Penn Nursing Science. A reinforcement phone call will be conducted one month later, and the session repeated at six months.
  Arms: Nurse-Led Face-to-Face Educational Intervention

SUMMARY:
Heart failure is a chronic condition that can lead to frequent hospitalizations and reduced quality of life. This study aims to evaluate whether a nurse-led, face-to-face educational intervention can improve clinical stability, treatment compliance, and self-care behaviors among patients with heart failure after hospital discharge. Participants will be randomly assigned to either the intervention group, receiving a structured 30-minute educational session using the teach-back method, or the control group, receiving standard follow-up care. The primary outcome is clinical stability at three months, assessed using the Heart Failure Somatic Perception Scale. Secondary outcomes include self-care and medication compliance measured up to 12 months. The study will be conducted at the ASST di Lodi Heart Failure Clinic in Italy and is expected to last three years.

DETAILED DESCRIPTION:
Heart failure (HF) is a progressive chronic condition associated with high rates of readmission, mortality, and impaired quality of life. Adherence to therapy and self-care behaviors play a key role in maintaining clinical stability, yet many patients struggle to apply recommended management strategies after hospital discharge.

This randomized controlled trial (EDUCATE study) aims to assess the effectiveness of a nurse-led, face-to-face educational intervention on clinical stability, treatment compliance, and self-care in patients with HF during the post-discharge period. The intervention consists of a 30-minute educational session conducted by trained nurses during the first outpatient cardiology visit, approximately 30 days after discharge. The session includes symptom assessment, individualized education using the teach-back method, and delivery of educational materials from Penn Nursing Science. A follow-up reinforcement phone call will be made one month later, and the educational session will be repeated at six months.

Participants will be randomly assigned (1:1) to either the intervention or control group. The control group will receive standard follow-up care, including monthly telephone contacts to support medication adherence and symptom monitoring. The primary outcome is clinical stability at three months, measured by the Heart Failure Somatic Perception Scale. Secondary outcomes include self-care (Self-Care of Heart Failure Index 7.2) and medication compliance (Morisky 4-item Scale), assessed at 3, 6, 9, and 12 months.

The study will be conducted at the Heart Failure Clinic of ASST di Lodi, Italy, with an anticipated enrollment of 118 participants. The total study duration is 36 months, including 24 months of recruitment and 12 months of follow-up for the last enrolled participant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospital discharge from the Cardiology Unit of Lodi Hospital with a diagnosis of heart failure according to international guidelines
* NYHA functional class II-IV assigned at discharge
* First outpatient cardiology visit scheduled 30 (±15) days after hospital discharge
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Severe cognitive impairment (Six Item Screener score 0-3)
* Admission from a unit other than the Cardiology Department of Lodi Hospital
* NYHA class I
* First cardiology visit scheduled <30 or >45 days after discharge
* Previous enrollment or follow-up in any Heart Failure Clinic
* Acute coronary event within the previous 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Stability at 3 Months | 3 months after the first outpatient cardiology visit.
  Clinical stability will be assessed using the Heart Failure Somatic Perception Scale (HFSPS). The scale measures symptom perception in heart failure. A difference of at least 7 points between intervention and control groups (favoring the intervention) is hypothesized.

SECONDARY OUTCOMES:
Self-Care Lavels | 3, 6, 9, and 12 months after the first outpatient cardiology visit
  Self-care behaviors will be assessed using the Self-Care of Heart Failure Index version 7.2 (SCHFI 7.2). Higher scores indicate better self-care; scores >70 are considered adequate.
Medication Compliance | 3, 6, 9, and 12 months after the first outpatient cardiology visit
  Medication adherence will be measured with the 4-item Morisky Scale. A total score of 4 indicates high adherence. The proportion of participants reporting full adherence ("No" to all items) will be compared between groups.

OTHER OUTCOMES:
Health-Related Quality of Life | 3, 6, 9, and 12 months after the first outpatient cardiology visit
  Health-related quality of life will be measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ). Higher scores indicate better perceived quality of life and lower symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Greta Ghizzardi, Ph.D., Principal Investigator — Azienda Socio Sanitaria Territoriale di Lodi
Locations (1):
- Azienda Socio Sanitaria Territoriale di Lodi, Lodi, Lodi, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves clinical data collected within a single institution and is subject to privacy and data protection regulations under the EU General Data Protection Regulation (GDPR). Only aggregated, anonymized results will be made available in scientific publications or presentations.

REFERENCES:
- [Background] Centrella-Nigro AM, Alexander C. Using the Teach-Back Method in Patient Education to Improve Patient Satisfaction. J Contin Educ Nurs. 2017 Jan 1;48(1):47-52. doi: 10.3928/00220124-20170110-10. PMID 28099678
- [Background] Alpert CM, Smith MA, Hummel SL, Hummel EK. Symptom burden in heart failure: assessment, impact on outcomes, and management. Heart Fail Rev. 2017 Jan;22(1):25-39. doi: 10.1007/s10741-016-9581-4. PMID 27592330
- [Background] Riegel B, Dickson VV, Faulkner KM. The Situation-Specific Theory of Heart Failure Self-Care: Revised and Updated. J Cardiovasc Nurs. 2016 May-Jun;31(3):226-35. doi: 10.1097/JCN.0000000000000244. PMID 25774844
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827